CLINICAL TRIAL: NCT01734447
Title: Discontinued Administration (6 Months a Year) of Growth Hormone to Children With Very Short Stature and Having Suffered From Intrauterine Growth Retardation: Safety and Effect on Growth of Long-term Therapy
Brief Title: Long Term Effect of Somatropin in Subjects With Intrauterine Growth Retardation
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GHRETARD/F/2/F
Record Dates: First submitted 2012-11-22; First posted 2012-11-27 (Estimated); Last update posted 2017-02-28 (Actual); Status verified 2017-02

CONDITIONS: Foetal Growth Problem; Small for Gestational Age
MeSH Terms: interventions — Human Growth Hormone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1.2, continuous treatment (Experimental)
  Interventions: Drug: somatropin
- 1.2, non-continuous treatment (Experimental)
  Interventions: Drug: somatropin
- 2.4, non-continuous treatment (Experimental)
  Interventions: Drug: somatropin

INTERVENTIONS:
Drug: somatropin — 1.2 IU/kg/week, one injection per day, in six days out of seven days, for 12 months
  Arms: 1.2, continuous treatment
Drug: somatropin — 1.2 IU/kg/week, one injection per day, in six days out of seven days, for 6 months out of 12 months (i.e. alternating periods of 6 months of treatment and non-treatment, respectively)
  Arms: 1.2, non-continuous treatment
Drug: somatropin — 2.4 IU/kg/week, one injection per day, in six days out of seven days, for 6 months out of 12 months (i.e. alternating periods of 6 months of treatment and non-treatment, respectively)
  Arms: 2.4, non-continuous treatment

SUMMARY:
This trial is conducted in Europe. The aim of this trial is to assess the safety of long-term growth hormone treatment in growth-retarded children with intrauterine growth retardation (IUGR) enrolled in trial GHRETARD/F/1/F.

ELIGIBILITY:
Inclusion Criteria:

* Patients born with IUGR enrolled in trial GHRETARD/F/1/F
* Bone age below 14 years in boys and 12 years in girls

Exclusion Criteria:

* Bone age above 14 years in boys and 12 years in girls

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2000-04-30 (Actual); Primary Completion 2003-04-30 (Actual); Study Completion 2003-04-30 (Actual)

PRIMARY OUTCOMES:
Glucose tolerance as assessed by hyperglycaemia induced by oral ingestion

SECONDARY OUTCOMES:
Bone Age determined according to Greulich and Pyle method and measured on the left hand X-ray
Pubertal development, assessed according to Tanner method
Height velocity
Final height
Number of Adverse Events

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (1):
- Novo Nordisk Investigational Site, Paris, France

REFERENCES:
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com